CLINICAL TRIAL: NCT00000768
Title: A Randomized Comparative Pharmacokinetic Study of Oral Ganciclovir After Treatment With Intravenous Ganciclovir for Cytomegalovirus Gastrointestinal Disease in AIDS Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 183; 11158 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Colitis; HIV Infections
Keywords: Intestinal Absorption; Ganciclovir; Drug Therapy, Combination; Cytomegalovirus Infections; Colitis; Administration, Oral; Acquired Immunodeficiency Syndrome; Biological Availability; Glutamic Acid
MeSH Terms: conditions — Colitis; HIV Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Glutamic acid hydrochloride
Drug: Ganciclovir

SUMMARY:
To determine the oral bioavailability of three dose levels of oral ganciclovir given with and without glutamic acid hydrochloride in patients with cytomegalovirus (CMV) GI disease, and to compare the bioavailability of these regimens to that of standard intravenous (IV) ganciclovir.

Long-term ganciclovir maintenance therapy has been recommended for CMV colitis or esophagitis following induction treatment. Oral ganciclovir is a likely candidate for maintenance because of its possible therapeutic value and ease of administration, but an optimum dose has not been determined. Since oral ganciclovir has a low bioavailability and is more soluble in an acid pH environment, the addition of glutamic acid hydrochloride may enhance gastrointestinal absorption of this drug.

DETAILED DESCRIPTION:
Long-term ganciclovir maintenance therapy has been recommended for CMV colitis or esophagitis following induction treatment. Oral ganciclovir is a likely candidate for maintenance because of its possible therapeutic value and ease of administration, but an optimum dose has not been determined. Since oral ganciclovir has a low bioavailability and is more soluble in an acid pH environment, the addition of glutamic acid hydrochloride may enhance gastrointestinal absorption of this drug.

All patients receive an induction regimen of IV ganciclovir administered twice daily for 21 to 42 (Per Amendment 3/4/95) days. A permanent venous catheter is implanted for the induction therapy. If clinically improved following induction, patients are then randomized to receive one of three doses of oral ganciclovir, given first without and then with oral glutamic acid hydrochloride, every 8 hours until they reach a steady state. PER AMENDMENT 3/14/95: After subjects have reached steady state with oral ganciclovir and glutamic acid hydrochloride then PK samples will be taken. Subjects will continue the dosing regimen they were assigned to (glutamic acid hydrochloride will be added if it resulted in at least 33% increased bioavailability) for up to 12 months or until relapse of CMV GI disease is documented. Subjects will be followed at monthly intervals for safety evaluation and for evidence of CMV GI relapse. Subjects who have clinical symptoms of relapse will undergo repeat endoscopy or colonoscopy to document the relapse.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis.

Allowed:

* Antiretroviral therapy during induction and pharmacokinetic part of study, provided patient remains on the same antiretroviral therapy for the duration of the study.
* Chemotherapy for Kaposi's sarcoma, provided patient is hematologically stable for at least 30 days prior to study entry.
* Recombinant human erythropoietin.
* GM-CSF and G-CSF.
* Other medications necessary for patient's welfare, at the physician's discretion.

Patients must have:

* HIV infection.
* Biopsy-proven cytomegalovirus (CMV) colitis.
* Life expectancy of at least 3 months.
* No active AIDS-defining opportunistic infection requiring therapy that is known to cause nephrotoxicity or myelosuppression.

NOTE:

* Kaposi's sarcoma is permitted if patients are hematologically stable for at least 30 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Other etiologies for diarrhea identified at study entry.

PER AMENDMENT 3/14/95:

* For subjects who have diarrhea - no other etiologies for diarrhea identified within 6 weeks of enrollment.
* Known hypersensitivity to study drugs.
* CMV retinitis.

Concurrent Medication:

Excluded:

* Acyclovir or probenecid (PER AMENDMENT 3/14/95).
* Immunomodulators.
* Biologic response modifiers (other than GM-CSF or G-CSF).
* Investigational agents, with the exception of treatment IND drugs.
* Antacids.
* H2 blockers.
* Proton pump inhibitors.
* Foscarnet during induction and pharmacokinetic part of study.
* Intravenous CMV retinitis maintenance therapy (including ganciclovir) during pharmacokinetic part of study.
* Nephrotoxic agents.

Prior Medication:

Excluded within 14 days prior to study entry:

* Immunomodulators.
* Biologic response modifiers (other than GM-CSF or G-CSF).
* Investigational agents, with the exception of treatment IND drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Study Completion 1998-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobson M, Study Chair; Dieterich D, Study Chair; Kotler D, Study Chair; Laine L, Study Chair; Kumar P, Study Chair
Locations (5):
- United States (5):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Ucsf Aids Crs, San Francisco, California
  - Washington U CRS, St Louis, Missouri
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio

REFERENCES:
- [Background] Dieterich DT, Kotler DP, Busch DF, Crumpacker C, Du Mond C, Dearmand B, Buhles W. Ganciclovir treatment of cytomegalovirus colitis in AIDS: a randomized, double-blind, placebo-controlled multicenter study. J Infect Dis. 1993 Feb;167(2):278-82. doi: 10.1093/infdis/167.2.278. PMID 8380610